CLINICAL TRIAL: NCT03746990
Title: Evaluation of Degree of Enamel Fluorosis in Children of Tobruk and Kufra Regions in Libya
Brief Title: Presence of Enamel Fluorosis in Libyan Children
Status: Completed | Type: Observational
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, ASSISTANT PROFESSOR, Ajman University
Other Study IDs: 6/24/17
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Dental Fluorosis
Keywords: fluoride; mottling; libya; fluorosis
MeSH Terms: conditions — Fluorosis, Dental; Fluoride Poisoning

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational: Total of 2015 Libyan school children aged 7 to 16 years, from urban (Tobruk) and rural (Kufra) areas were included in the main study. The children were of almost equal number of both sexes from each age group (table-I) .The total of 1935 children were examined for enamel fluorosis

SUMMARY:
Fluorosis is caused by hypomineralization in the enamel due to increased fluoride ingestion during early childhood (Cawson.1, Wong et al. 2, and Sudhir 3). A considerable amount of evidence has been reported over the years, which has shown that presence of fluoride ions at up to one part per million in public water supply has reduced the prevalence of teeth decayed with minimal chance of dental fluorosis. The WHO recognized these facts by its resolution in 1969 4 and 1975 5, which stated that water fluoridation, where applicable, should be the cornerstone of any national policy of caries prevention

DETAILED DESCRIPTION:
The optimal concentration is defined as that which gives maximal protection against dental caries, with minimal clinically observable dental fluorosis (Dunning 7). This level is determined according to the climate and the resultant drinking habits (Newborn 6). Cawson 1 stated that mottling of enamel is the most frequently seen and most reliable sign of excessive quantities of fluoride in the drinking water. Dean 8 concluded that a fluoride level of above 1ppm does not significantly reduce caries beyond the optimal effect of 1ppm.

Different classifications have been introduce to score dental fluorosis. (Dean 9, Al -Alousi 10, Thylstrup & Fejerskov 11, (Fejerskov, 12). and the DDE index by FDI 1982). Aira Sabokseir 13, concluded, fluorosis indices, if used alone, could result in misdiagnosis of dental fluorosis and information about adverse health-related conditions linked to DDEs (Developmental Defects of Enamel) at specific positions on teeth could help to differentiate between genuine fluorosis and fluorosis-resembling defects.Various figures for mouth prevalence of enamel fluorosis have been reported by different investigators. 39.2% by Al-Alousi 10, for Welsh children, 32% by Akpata 14 for Nigerian children. Using the DDE index of the FDI (1982), Al alousi 10 defective enamel of 48.9% in children from south Wales. In England,Tabari 15 found the prevalence of fluorosis was 54% in the fluoridated area and 23% in the fluoride-deficient area. In Iran the prevalence of fluorosis was 61% (Azami-Aghdash et al., 16).

ELIGIBILITY:
Inclusion Criteria:

* Libyan children born and lived in the same area. 2. Limited to incisors only.

Exclusion Criteria:

* Non- Libyan children. 2. Children who born or lived outside the study areas. 3. Incisors with class II fracture (Ellis type 1970) or crowned

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study is part of a cross - sectional investigation of aspects of dental health in rural and urban Libyan school children. Total of 2015 Libyan school children aged 7 to 16 years, from urban (Tobruk) and rural (Kufra) areas were included in the main study. The children were of almost equal number of both sexes from each age group (table-I) .The total of 1935 children were examined for enamel fluorosis, the remaining, eighty children were excluded because they failed to meet inclusive criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1935 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Grading of mottling | From baseline to 5 months
  If there was fluorosis, the tooth or teeth were diagnosed as having fluorosis and coded according to the method produced by Al- Alousi 10, as follows A. White areas less than 2mm in diameter. B. White areas of or greater than 2mm in diameter. C. Colored (brown) areas less than 2mm in diameter, irrespective of there being any white areas.
  D. Colored (brown) areas of or greater than 2mm in dimeter, irrespective of there being any white area.
  E. Horizontal white lines irrespective of there being any white, non-linear areas.
  F. Colored (brown) or hypo-plastic areas.

CONTACTS AND LOCATIONS:
Overall Officials: suleiman r ergieg, Phd, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No